CLINICAL TRIAL: NCT00438373
Title: Association of LH/HCG Receptor Expression and Retrieval Rates at Oocyte Pick up.
Brief Title: LH/HCG Receptor Expression and Retrieval Rates
Status: Suspended | Type: Observational
Sponsor: Aristotle University Of Thessaloniki (Other)
Collaborators: University of Athens (Other)
Responsible Party: Principal Investigator, E.M. Kolibianakis, Professor, Aristotle University Of Thessaloniki
Other Study IDs: UHR-1
Record Dates: First submitted 2007-02-21; First posted 2007-02-22 (Estimated); Last update posted 2015-02-26 (Estimated); Status verified 2015-02

CONDITIONS: Subfertility
Keywords: Subfertility, Luteinizing hormone, receptor
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The purpose of this study is to evaluate if there is an association between the serum LH receptor expression on the day of hCG administration or the day of oocyte retrieval and the retrieval rates at oocyte pick up

DETAILED DESCRIPTION:
The purpose of this study is to evaluate if there is an association between the serum LH receptor expression on the day of hCG or the day of oocyte retrieval and the retrieval rates at oocyte pick up.

For this purpose, m-RNA copy numbers will be assessed in the blood serum of patients undergoing ovarian stimulation for IVF on different days.

Furthermore, detailed ultrasound scans will be perfomed, as well as assesment of hormonal levels during ovarian stimulation.

ELIGIBILITY:
Inclusion criteria:

* Age <39 years,
* Body mass index (BMI) between 18 and 29 kg/m2,
* Presence of both ovaries,
* FSH levels <10 IU/l.

Exclusion criteria:

* Endometriomas,
* Polycystic ovarian syndrome.

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: infertile patients undergoing assisted reproduction tratment
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2007-01; Primary Completion 2016-01 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
LH/hCG receptor expression | at oocyte retrieval

CONTACTS AND LOCATIONS:
Overall Officials: Basil C Tarlatzis, MD, PhD, Study Director — Unit of Human Reproduction, 1st Department of Obs & Gyne, Aristotle University of Thessaloniki, Papageorgiou Hospital, Greece
Locations (1):
- Unit of Human Reproduction, 1st Department of Obstetrics & Gynecology, AUTH, Papageorgiou Hospital, Thessaloniki, Greece

REFERENCES:
- [Background] Patsoula E, Loutradis D, Drakakis P, Michalas L, Bletsa R, Michalas S. Messenger RNA expression for the follicle-stimulating hormone receptor and luteinizing hormone receptor in human oocytes and preimplantation-stage embryos. Fertil Steril. 2003 May;79(5):1187-93. doi: 10.1016/s0015-0282(03)00071-2. PMID 12738515
- [Background] Patsoula E, Loutradis D, Drakakis P, Kallianidis K, Bletsa R, Michalas S. Expression of mRNA for the LH and FSH receptors in mouse oocytes and preimplantation embryos. Reproduction. 2001 Mar;121(3):455-61. doi: 10.1530/rep.0.1210455. PMID 11226072